CLINICAL TRIAL: NCT06021184
Title: Impact of the Approximate Dose-Equivalent of Fibrinogen-to-Erythrocyte Suspension (ADEFES) Ratio on Mortality and Functional Outcomes in Patients with Major Intraoperative Bleeding- a Prospective Observational Trial (ADEFES Trial)
Brief Title: "ADE Fibrinogen/RBC" Ratio on Mortality and Outcome in Massive Transfusion Patients
Acronym: ADEFES
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Istanbul University (Other); Ondokuz Mayıs University (Other); Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other); Kanuni Sultan Suleyman Training and Research Hospital (Other); Saglik Bilimleri Universitesi (Other); Sakarya University (Other); Acibadem Atakent University Hospital (Other); Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ADEFES
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Massive Transfusion; Bleeding During/following Surgery
Keywords: massive transfusion; fibrinogen; fresh frozen plasma; red blood cell; cryoprecipitate; erythrocyte suspension; bleeding surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our study focuses on the transfusion of blood and blood products in cases of major bleeding, including massive transfusion scenarios where repeated doses of packed red blood cells (PRBC), fresh frozen plasma (FFP), cryoprecipitate, and fibrinogen concentrate are administered. Each of these blood products contains varying amounts of fibrinogen. Previous research has explored formulas to enhance outcomes by examining transfusion ratios such as FFP/ES, ES/platelet, and FFP/ES/platelet.

Building on this, our hypothesis is that increasing the total fibrinogen content provided within a short period of time from the beginning of major bleeding reduces mortality and morbidity. To standardize the fibrinogen amounts from different sources under a single pool, we developed a formula that equalizes the fibrinogen content across these products. Using the below formula, we aim to investigate the impact of the overall ADEF/ES ratio on mortality and functional outcomes in major bleeding.

Approximate Dose-Equivalent for Fibrinogen (ADE): 1 gram of fibrinogen = 5 units of cryoprecipitate = 1.5 units of FFP, evaluated as total grams of fibrinogen.

DETAILED DESCRIPTION:
Massive transfusion, defined as the transfusion of total body blood volume (10 units of erythrocyte suspension or 8 units and above in some definitions) or more within 24 hours, remains one of the greatest challenges for the anesthetist. Despite all the medical advances, in cardiac surgery, obstetric surgery, trauma-orthopedic surgery, neurosurgery, major gastrointestinal-genitor-urinary system surgeries, which are among the major bleeding surgeries, massive hemorrhage continues to be an important mortality and morbidity factor. In addition to major surgeries with known expected bleeding, massive transfusion requirement may arise with any undesirable intraoperative event. While the process is easier to manage with proper preparation and an organized procedure in expected bleeding, a chaotic response may be encountered in unexpected situations. Special protocols for each division have been developed by clinicians to manage this critical process, and work continues on these protocols to improve the outcome.

Massive bleeding management mainly focuses on transfusion and fluid resuscitation. Regardless of the situation requiring massive transfusion, the goals of treatment in massive bleeding are to maintain organ perfusion pressure and oxygen delivery, immediately stop bleeding and coagulopathy. While these goals can be achieved through resuscitation with blood products and surgical intervention, the triad of hypothermia, acidosis, and coagulopathy that occurs with the process contributes to increased morbidity and mortality in such scenarios.

The literature on major bleeding from trauma has highlighted some issues contributed to improved clinical outcomes such as, damage-controlled resuscitation, including timely initiation of transfusion, early use of clotting factors, minimizing the use of crystalloids. The landmark PROPPR study found that in the resuscitation of trauma patients, a 1:1:1 ratio of FFP:platelet:ES transfusion during massive bleeding resulted in hemostasis in a greater number of patients (86% versus 78%) compared to a 1:1:2 ratio, additionally, they found fewer deaths from bleeding within 24 hours (14.6% versus 9.2%). However, no significant difference was found in 24-hour or 30-day overall mortality. In a systematic review evaluating retrospective data on transfusions for obstetric bleeding, it was shown that the amount of FFP administered was greater than the amount of ES. Since the mortality rate from massive obstetric hemorrhage is lower than that of traumatic hemorrhage, it is difficult to prospectively evaluate the effects of massive transfusion. This review recommends a FFP/ES ratio of ≥1, with the results of all retrospective studies described on transfusions for obstetric hemorrhage. Studies in cardiac surgery also suggest that higher rates of FFP/ES transfusion are associated with better outcomes in patients with massive bleeding.

In general, the high ratio of transfused FFP to ES in bleeding surgeries requiring massive transfusion has been associated with positive results. FFP contains all coagulation factors and fibrinogen, as well as restoring the volume deficit that occurs with major bleeding, which reduces the crystalloid requirement and prevents extra dilution of coagulation factors. Fibrinogen is the clotting factor whose level drops the fastest during bleeding. Fibrinogen is a unique coagulation building block that plays a role in both primary and secondary hemostasis. Based on the results of the RETIC trial, the effectiveness of fibrinogen supplementation in limiting blood loss appears to be strongly dependent on timing of fibrinogen administration and increasing levels above 200 mg·dL-1. The 5th Edition of the European Guidelines for the Management of Major Posttraumatic Hemorrhage and Coagulopathy recommends early and repeated monitoring of fibrinogen concentrations and/or polymerization and rapid correction of deficiencies. Accordingly, 3-4 g of fibrinogen concentrate or 15-20 units of cryoprecipitate is recommended as an initial dose in massive bleeding. While RETIC stands out as a randomized controlled prospective study on the role of fibrinogen in massive transfusion in trauma patients, there are few cardiac and transplantation surgery studies in various types of research. Regardless of the cause, early restoration of fibrinogen levels in case of massive bleeding reduces transfusion requirement by preventing ongoing bleeding. In the FIBRES study, which evaluated the efficacy of fibrinogen concentrate in cardiac surgery patients with bleeding, it was emphasized that fibrinogen concentrate was not inferior to cryoprecipitate, easy to apply, and a predictable robust effect. Further it is hypothesized that early replacement of fibrinogen in severely injured trauma patients may improve outcomes. However, there is little evidence to support this and, in addition, little evidence to support or refute the effects of cryoprecipitate or fibrinogen concentrate for fibrinogen replacement. Fibrinogen supplementation as cryoprecipitate within the first 90 minutes of major bleeding was considered feasable in a randomized controlled trial. As a matter of fact, in the E-FIT 1 study conducted with a very small number of patients, it was found that it is not effective to administer fibrinogen in the first 45 minutes. On the other hand, there is not only fibrinogen in the scene, results of the FIIRST 2 study comparing the use of combinations of fibrinogen concentrate and prothrombin complex concentrate (PCC) in hemorrhagic trauma patients are also eagerly awaited.

Ideally, fibrinogen concentrate and/or cryoprecipitate are used in fibrinogen replacement, and FFP is used as a weaker fibrinogen source. During massive transfusion, repeated doses of FFP/cryoprecipitate/fibrinogen concentrate are used. All of these blood products have different amounts of fibrinogen content. In many previous studies, the formula for improving the results was investigated by looking at transfusion rates such as FFP/ES, ES/platelet, FFP/ES/Platelet. In the light of this information, our hypothesis is that mortality and morbidity can be reduced with a high rate of total fibrinogen from various sources. In order to combine the fibrinogen amounts from different sources under a single name, we determined an equalization according to the fibrinogen amounts they contain. In accordance with this formula, it was considered to investigate the effect of the overall ADEF/ES ratio on mortality and outcome in massive transfusion cases that fit the definitions.

The primary aim of this study to determine the effect of the ratio of total fibrinogen to erythrocyte suspension (ADE Fibrinogen/ES) transfused at 24 hours on the composite outcome, which includes 30-day all-cause mortality, bleeding-specific mortality, and the Katz index of independence in activities of daily living (scored 0, 1, 2- i.e. extremely dependent to highly dependent).

The secondary aim of this study to determine the relationship of ADEF/ES ratio with other parameters:

* Postoperative 24-hour and 3-month all-cause and bleeding specific mortality
* Morbidity(>90 day) Morbidity defined as events continuing after 90 days (ICD code 9)

  * thrombotic event (DVT, Pulmonary Embolism, DIC)
  * respiratory event (ventilator-associated pneumonia, other surgery-related respiratory complications)
  * ischemic event (Myocardial infarction, TIA, Cerebrovascular accident)
  * infection (sepsis, surgical site infection, any drug-resistant infection)
  * permanent kidney damage
* Mortality predictors Mortality predictors as defined ;
* Age
* Gender
* ASA score
* Glasgow coma scale
* Charlson Comorbidity index
* Euroscore II
* TASH score
* Shock index
* ISTH (International Society on Thrombosis and Haemostasis) score
* ISS score
* AC SURGICAL RISK CALCULATOR
* History of antiplatelet-anticoagulant and ACEI or ARBs drug use
* Emergency surgery
* Temperature
* Surgery specific details (Type of surgery, Duration of surgery periods, cement use etc]
* Intraoperative Vasopressor-inotropic medicine Requirement
* Laboratory data over time

  - when statistic testing mortality the data will be adjusted for these predicting/contributing factors
* Complications Complications as defined;

  --- Cardiac complications
* Arrest
* New developed unstable Arrhythmia
* MI
* KKY
* Aortic dissection

  --- Kidney complications
* AKI I/II/III/IV (defined by KDIGO Criteria)
* CRRT (temporary)
* Continuous dialysis/CRF

  --- Lung complications
* Pulmonary edema
* Pneumothorax
* Pleural effusion
* ARDS/respiratory failure
* Bronchospasm
* Aspiration pneumonitis

  --- Neurological complications
* Ischemic cerebral events
* Hemorrhagic cerebral events (non-traumatic)
* Permanent sequelae
* TIA
* Seizure

  --- Infective complications
* Pneumonia
* Mediastinitis
* Meningitis
* Urinary tract infection
* Wound site infection (Surgical Site Infections)
* Catheter location infection
* Sepsis

  --- Thrombotic complications
* Deep vein thrombosis
* Pulmonary embolism
* Mesentery thromboembolism
* Stroke
* Other

  * MODS/SIRS
  * MT Complications
* Hematological Complications

  * Hemolytic rxns (Acute/delayed)
  * Febrile non-hemolytic reactions
  * DIC
  * Allergic reactions
  * TRALI (transfusion related acute lung injury)
  * TRAHI (transfusion related acute hepatic injury)
  * TACO (transfusion assoc. circulatory overload)
* Abdominal compartment syndrome

  --- Ischemic hepatitis, shock liver
* Length of stay in the ICU Length of stay in the hospital
* Functional state at discharge (can perform daily activities, can perform daily activities with assistance, completely in need of help)
* All cause and bleeding specific mortality- Surgery specific postoperative 24-hour, 30 day and 3-month
* Katz index of independence in activities of daily living (0,1,2 bad and 5,6 good scores)- Surgery specific postoperative 24-hour, 30 day and 3-month
* Tranexamic acid use and mortality relationship
* Initial(admission) plasma fibrinogen level and amount of bleeding Initial(admission) plasma fibrinogen level and amount of ADEF

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18
2. Surgical patients who received ''Transfusion of ≥ 4 U ESs and at least one fibrinogen-containing product (FFP, fibrinogen concentrate, cryoprecipitate) within 24 hours''
3. Elective or emergency surgical procedures with major bleeding. Major bleeding surgeries; cardiovascular and thoracic surgery, obstetric-gynecologic surgery, orthopedics/trauma surgery, neurosurgery, transplantation and major ENT-GIS-GUS surgeries.
4. Informed Consent
5. Undergoing surgery within 24 hours of massive blood transfusion

Exclusion Criteria

1. Death before massive transfusion
2. Death during massive transfusion
3. Patients whose perioperative bleeding and transfusion data cannot be accessed in detail
4. Patients with missing data or non-compliance with study protocol
5. Patients who have zero ADEF/ES ratio

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who received at least 4 unite RBC transfusion and a fibrinogen containing product
Sampling Method: Probability Sample
Enrollment: 1679 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite score of any one of the following events occurring 30 days within the beginning of transfusion: | From enrollment (beginning of transfusion for surgical bleeding) to the end of 30 days
  (1) 30-day all-cause mortality, (2) bleeding-specific mortality, (3) the Katz index of independence in activities of daily living.
  To determine the effect of the ratio of total fibrinogen to erythrocyte suspension (ADE Fibrinogen/ES) transfused at 24 hours on the composite outcome, which includes 30-day all-cause mortality, bleeding-specific mortality, and the Katz index of independence in activities of daily living (scored 0, 1, 2) i.e. extremely dependent to highly dependent).

SECONDARY OUTCOMES:
Postoperative 24-hour all-cause and bleeding specific mortality | From enrollment (beginning of transfusion for surgical bleeding) to the end of 24 hour
  To determine the ADEF/ES ratio relationship with postoperative 24-hour all-cause and bleeding-specific mortality.
Postoperative 3-month all-cause and bleeding specific mortality | From enrollment (beginning of transfusion for surgical bleeding) to the end of 3 month
  To determine the ADEF/ES ratio relationship with postoperative 3-month all-cause and bleeding specific mortality.
Morbidity(>90 day) | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with morbidity continuing after 90 days.
  Morbidity defined as events continuing after 90 days (ICD code 9)
  * thrombotic event
  * respiratory event
  * ischemic event
  * infection
  * permanent kidney damage
Mortality predictors | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with below parameters.
  * Age
  * Gender
  * ASA score
  * Glasgow coma scale
  * Charlson Comorbidity index
  * Euroscore II
  * TASH score
  * Shock index
  * ISTH (International Society on Thrombosis and Haemostasis) score
  * ISS score
  * AC SURGICAL RISK CALCULATOR
  * History of antiplatelet-anticoagulant and ACEI or ARBs drug use
  * Emergency surgery
  * Temperature
  * Surgery specific details (Type of surgery, Duration of surgery periods, cement use etc]
  * Intraoperative Vasopressor-inotropic medicine Requirement
  * Laboratory data over time
Cardiac complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * Arrest
  * New developed unstable Arrhythmia
  * MI
  * KKY
  * Aortic dissection
Kidney complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * AKI I/II/III/IV (defined by KDIGO Criteria)
  * CRRT (temporary)
  * Continuous dialysis/CRF
Lung complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * Pulmonary edema
  * Pneumothorax
  * Pleural effusion
  * ARDS/respiratory failure
  * Bronchospasm
  * Aspiration pneumonitis
Neurological complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * Ischemic cerebral events
  * Hemorrhagic cerebral events (non-traumatic)
  * Permanent sequelae
  * TIA
  * Seizure
Infective complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * Pneumonia
  * Mediastinitis
  * Meningitis
  * Urinary tract infection
  * Wound site infection (Surgical Site Infections)
  * Catheter location infection
  * Sepsis
Thrombotic complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * Deep vein thrombosis
  * Pulmonary embolism
  * Mesentary thromboembolism
  * Stroke
  * Other
MODS | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the MODS (multiple organ dysfunction syndrome) in patients
SIRS | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the systemic inflammatory response syndrome (SIRS)
Massive Transfusion Complications | 90 days after registration (from the start of transfusion for surgical bleeding)
  To determine the ADEF/ES ratio relationship with the below definition
  * Hematological Complications Hemolytic reaction (Acute/delayed) Febrile non-hemolytic reactions DIC (Disseminated Intravascular Coagulation) Allergic reactions TRALI (transfusion-related acute lung injury) TRAHI (transfusion-related acute hepatic injury) TACO (transfusion assoc. circulatory overload)
  * Abdominal compartment syndrome
  * Ischemic hepatitis, shocked liver
ICU (intensive care unit) stay | From enrollment (beginning of transfusion for surgical bleeding) to the end of 3 month
  The patient's total ICU (intensive care unit) stay will be recorded.
Total length of hospital stay | From enrollment (beginning of transfusion for surgical bleeding) to the end of 3 month
  The total length of patient's hospital stay will be recorded.
Functional state at discharge | From enrollment (beginning of transfusion for surgical bleeding) to the end of 3 month
  To determine the ADEF/ES ratio relationship with Functional state at discharge (can perform daily activities, can perform daily activities with assistance, completely in need of help)
The Katz Index of Independence in activities of daily living tool | From enrollment (beginning of transfusion for surgical bleeding) to the end of 3 month
  To determine the ADEF/ES ratio relationship with Katz score. Objective assessment is made by the KATZ index of independence of activities of daily living. The Katz index measures six self-care tasks including; bathing, dressing, toileting, transferring, maintaining continence, and feeding using a dichotomous rating. Katz index of independence in activities of daily living (0,1,2 bad and 5,6 good scores). Surgery specific postoperative 24-hour, 30 day and 3-month
Tranexamic acid | From enrollment (beginning of transfusion for surgical bleeding) to the end of 3 month
  Tranexamic acid use and mortality relationship.
Initial (admission) plasma fibrinogen level | Beginning of transfusion for surgical bleeding
  Initial (admission) plasma fibrinogen level will be recorded. To determine the relationship between initial (admission) plasma fibrinogen level and amount of bleeding.
Plasma fibrinogen level initial (admission) | Beginning of transfusion for surgical bleeding
  Initial (admission) plasma fibrinogen level will be recorded. To determine the relationship between initial (admission) plasma fibrinogen level and amount of ADEF.

CONTACTS AND LOCATIONS:
Overall Officials: Kemalettin Koltka, Prof, Study Chair — Istanbul University
Locations (1):
- Ankara Bilkent city hospital, Ankara, çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demir ZA, Kavak Akelma F, Akca O, Koltka K, Dincer B, Kocyigit M, Tuna AT, Sayin J, Yildirim Ar A, Kuvaki B, Aykut A, Sahin AS, Aydin Guzey N; ADEFES Investigators. Impact of fibrinogen-to-erythrocyte suspension ratio on mortality and functional outcomes in major perioperative bleeding (Approximate Dose-Equivalent of Fibrinogen-to-Erythrocyte Suspension (ADEFES) study): protocol for a prospective observational study. BMJ Open. 2025 Sep 16;15(9):e099044. doi: 10.1136/bmjopen-2025-099044. PMID 40962355